CLINICAL TRIAL: NCT01135797
Title: Retrospective Safety Survey In Patients Included In Phase I-II NV1FGF Clinical Trials
Brief Title: Retrospective Safety Survey In Patients Included In NV1FGF Clinical Trials
Acronym: TALISMAN S
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Other Study IDs: LTS11315
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients from phase I-II studies

SUMMARY:
The objective of this study is to collect retrospectively long term safety data in patients who have participated in the previous phase I-II trials conducted with the compound.

ELIGIBILITY:
Inclusion criteria:

* Patient randomized, treated and alive at the end of the phase I-II study participation, irrespective of their treatment group,
* Who signed the TALISMAN survey informed consent (or for deceased patients, the informed consent was signed the legal representative/family member as per national regulations - except in countries where Ethics Committee approval only is required for retrospective data collection).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in this observational study previously participated in one of the phase I-II studies for the compound
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Deaths | From the end of their participation in the phase I-II study until 36 months (+/- 3 months) after their first study drug intake
  Including all causes of deaths
Incidence of safety events of interest | From the end of their participation in the phase I-II study until 36 months (+/- 3 months) after their first study drug intake
  Safety events of interest when gene therapy is used i.e. development of any new/recurrent cancer, immunogenicity reactions

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom